CLINICAL TRIAL: NCT04393428
Title: Urinary Biomarkers (TIMP-2 and IGFBP7) for Early Diagnostic Assessment of Acute Kidney Injury in Patients With SARS-CoV-2 (COVID-19)
Brief Title: Urinary Biomarkers for AKI Diagnosis in Patients With SARS-CoV-2 (COVID-19)
Acronym: COVID-AKI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0294
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Renal Replacement Therapy; Acute Kidney Injury
Keywords: Acute Kidney Injury; SARS-CoV-2; Renal Replacement Therapy
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients with urinary samples: COVID-19 patients with urinary samples
  Interventions: Other: [TIMP-2]*[IGFBP-7]

INTERVENTIONS:
Other: [TIMP-2]*[IGFBP-7] — [TIMP-2]*[IGFBP-7] mesurement in urine sample relicates of COVID-19 patients admitted to the Montpellier University Hospital

SUMMARY:
Among patients with SARS-CoV-2 pneumonia, approximately 20% have an acute kidney injury (AKI) and 5% require renal replacement therapy. Occurrence of AKI in patients with COVID-19 is associated with increased morbidity and mortality. Early detection of patients at risk of AKI would allow to prevent onset or worsening of AKI. The aim of this study is to determine if urine biomarkers of renal tubular damage such as TIMP-2 and IGFBP7 could early identify patients with SARS-CoV-2 pneumonia at risk of developing AKI.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* COVID-19 confirmed by positive SARS-CoV-2 PCR
* at least one urine sample

Exclusion criteria:

* Persons under protection
* Paritcipation rejections

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients admitted to the Montpellier University Hospital with at least one rine sample drawn
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sensibility and specificity of urinary | Occurence of AKI 7 days after urinary biomarkers measurement
  Sensibility and specificity of urinary [TIMP-2]*[IGFBP-7] > 0,3 to predict AKI (KDIGO stage ≥ 1) in SARS-CoV-2 patients at day-7 after measurement

SECONDARY OUTCOMES:
Sensibility and specificity of urinary | Occurnce of AKI worsening, renal replacement therapy requirement or persistant AKI, 7 days after urinary biomarkers mesurement
  Sensibility and specificity of urinary [TIMP-2]*[IGFBP-7] > 0,3 to predict AKI worsening, renal replacement therapy requirement or persistant AKI

CONTACTS AND LOCATIONS:
Overall Officials: Romaric Larcher, MD, PharmD, MSc, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC